CLINICAL TRIAL: NCT03935594
Title: Use of Autologous Platelet-Rich Plasma to Treat Hypertrophic Burn Scars; A Randomized Controlled Double-Blinded Trial
Brief Title: Use of Autologous Platelet-Rich Plasma to Treat Hypertrophic Burn Scars
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Intervention causing discomfort to participants
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Salam Al Kassis, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #190170
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Hypertrophic Scar
Keywords: platelet rich plasma (PRP); hypertrophic scar; burn scar; tissue repair; vancouver scar scale (VSS); patient and observer scar assessment scale (POSAS)
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All patients meeting inclusion/exclusion criteria will be offered enrollment. Using a coin flip, patients will have a 50% chance of receiving PRP injection on the right half of the scar (as opposed to the left half). Multiple scar sites may be enrolled per patient, without limit.
Who Masked: Participant
Masking Description: Patients will be blinded to which halves of their scar are in either arm of the study. On each visit, before the patient is able to see the contents of syringes used for injection of either normal saline or platelet rich plasma, the syringes will be covered with a white sticker and labeled such that the provider knows which syringe has PRP vs normal saline but the patient does not (PRP is yellow and normal saline is clear). Depending on which side (left vs right) was assigned PRP vs normal saline, the appropriate area will be injected with 1mL/1sq-cm of PRP or normal saline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP injection right half (Experimental): The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the control half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL normal saline into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
  Interventions: Biological: PRP Injection; Drug: Saline Injection
- PRP injection left half (Experimental): The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the experimental half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL PRP into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
  Interventions: Biological: PRP Injection; Drug: Saline Injection

INTERVENTIONS:
Biological: PRP Injection — 1mL platelet rich plasma will be injected into each 1cm x 1cm area of scar tissue of the experimental half of the scar.
Drug: Saline Injection — 1mL NS will be injected into each 1cm x 1cm area of scar tissue of the control half of the scar.

SUMMARY:
Hypertrophic burn scars are experienced by more than 70% of burn victims. They are a major source of decreased quality of life in burn patients due to pain, decreased range of motion, and poor cosmetic appearance. Current treatment strategies (including fat grafting and laser resurfacing) are either highly invasive, prohibitively costly, or painful. Autologous Platelet Rich Plasma (PRP) does not require anesthesia, and is an inexpensive, safe, fast, and less painful alternative that has been recognized for its role in reducing scars associated with acne, among other things. While PRP has not been studied specifically in burn scars, there is sufficient theoretical and practical evidence that it will improve the appearance and feel of these debilitating scars, representing a large potential benefit for these patients with minimal associated risk.

DETAILED DESCRIPTION:
Severe burn injury is associated with hypertrophic scarring, which occurs in up to 70% of burn patients (Finnerty et al., 2016). Burn scars are particularly troublesome because they cause debilitating neuropathic pain and itch, joint contractures and stiffness that limit range of motion, inability to sweat, and physical disfigurement of cosmetically sensitive areas such as the hands and face.

Autologous platelet-rich plasma (PRP) is plasma with a higher concentration of platelets, and is prepared by drawing up a small amount of a patient's blood, centrifuging it, and collecting the platelet-rich layer. Many automated machines exist for doing this process. Platelets contain a multitude of growth factors and other small molecules that have been shown to promote wound healing and tissue regeneration in a variety of contexts. PRP, which is rich in these healing growth factors, has been studied extensively and has proved to be both a safe and effective treatment modality for a wide range of applications, including acne scars and hair loss (Elghblawi et al., 2018). It has been shown to be a safe and effective treatment for some types of surgical and traumatic scars, and has been safely applied to acute burn wounds where it has been shown to improve healing and subsequent scarring (Venter et al., 2016). Despite these known uses of PRP, its role in reducing the extent and severity of mature hypertrophic burn scars after they have already healed is notably lacking in the literature.

The purpose of this study is to assess whether intradermally-injected autologous platelet-rich plasma improves the size, texture, color, elasticity, contour, and neuropathic pain associated with mature burn scars.

Specific Aims:

1. Compare the effectiveness of intradermally-injected autologous platelet-rich plasma versus normal saline (NS) to improve burn scars, as measured by both clinician-reported (Vancouver scar scale; VSS) and patient-reported measures (Patient and Observer Scar Assessment Scale; POSAS).
2. Compare the effectiveness of intradermally-injected autologous platelet-rich plasma versus normal saline as a control to improve neuropathic pain associated with burn scars.
3. Understand the mechanism of action of PRP in improving burn scars via histological analysis of collagen content in the burn scar tissue biopsy specimens.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic burn scar present on trunk or abdomen

Exclusion Criteria:

* Initial burn injury less than 1 year old
* History of chemical or electrical burn
* Genetic or acquired conditions that severely affect systemic wound healing or collagen formation (vasculitis, diabetes, Ehlers-Danlos syndrome, radiation therapy to the scar site or use of immunosuppressive medications within the last year, active cancer)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2022-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galen Perdikis, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
All reasonable efforts will be made to keep a patient's protected health information (PHI) private and confidential. Electronic records will be stored in restricted access database (Redcap, Vanderbilt) open only to the study team or on sponsor electronic databases which are password protected.

REFERENCES:
- [Background] Cervelli V, Nicoli F, Spallone D, Verardi S, Sorge R, Nicoli M, Balzani A. Treatment of traumatic scars using fat grafts mixed with platelet-rich plasma, and resurfacing of skin with the 1540 nm nonablative laser. Clin Exp Dermatol. 2012 Jan;37(1):55-61. doi: 10.1111/j.1365-2230.2011.04199.x. PMID 22182435
- [Background] Prochazka V, Klosova H, Stetinsky J, Gumulec J, Vitkova K, Salounova D, Dvorackova J, Bielnikova H, Klement P, Levakova V, Ocelka T, Pavliska L, Kovanic P, Klement GL. Addition of platelet concentrate to dermo-epidermal skin graft in deep burn trauma reduces scarring and need for revision surgeries. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2014 Jun;158(2):242-58. doi: 10.5507/bp.2013.070. Epub 2013 Sep 27. PMID 24108222
- [Background] Ruiz A, Cuestas D, Garcia P, Quintero J, Forero Y, Galvis I, Velasquez O. Early intervention in scar management and cutaneous burns with autologous platelet-rich plasma. J Cosmet Dermatol. 2018 Dec;17(6):1194-1199. doi: 10.1111/jocd.12554. Epub 2018 Apr 22. PMID 29682893
- [Background] Asif M, Kanodia S, Singh K. Combined autologous platelet-rich plasma with microneedling verses microneedling with distilled water in the treatment of atrophic acne scars: a concurrent split-face study. J Cosmet Dermatol. 2016 Dec;15(4):434-443. doi: 10.1111/jocd.12207. Epub 2016 Jan 8. PMID 26748836
- [Background] Klosova H, Stetinsky J, Bryjova I, Hledik S, Klein L. Objective evaluation of the effect of autologous platelet concentrate on post-operative scarring in deep burns. Burns. 2013 Sep;39(6):1263-76. doi: 10.1016/j.burns.2013.01.020. Epub 2013 Mar 5. PMID 23481151

RESULTS

PARTICIPANT FLOW:
Groups:
- Scar Area (Control+Treated): The scar will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the control half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL normal saline into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  The area inside the experimental half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL PRP into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
Period: Overall Study
Arm/Group | Scar Area (Control+Treated)
Started | 3
PRP Treated | 3
Control | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Groups:
- Scar Area (Control + PRP): The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the control half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL normal saline or 1mL PRP into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
Arm/Group | Scar Area (Control + PRP)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Scar Assessment: POSAS at 2 Months
Description: Scar will be measured by Patient and Observer Scar Assessment Scale ( POSAS ) on both sides of the scar. POSAS score is an assessment of scar severity. The range is 6-60. 6=normal skin and 60= severely scarred skin.
Time Frame: 2 months
Population: We will report the POSAS median score of 3 participants at 2 months after injection.
  The initial plan was to recruit 40 participants and follow-up with them up to 6 months; however, the study was terminated at 2 months after the recruitment of 3 subjects only due to discomfort caused by the intervention.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Saline Injected Half: The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the control half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL normal saline into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
- PRP Injected Half: The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the experimental half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL PRP into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
  PRP Injection: 1mL platelet rich plasma will be injected into each 1cm x 1cm area of scar tissue of the experimental half of the scar.
Arm/Group | Saline Injected Half | PRP Injected Half
Number analyzed (Participants) | 3 | 3
score on a scale | 43 [26 to 43] | 39 [21 to 42]

2. Primary Outcome: Scar Assessment: VSS at 2 Months
Description: Scar will be measured by Vancouver Scar Scale (VSS) on both control half and experimental half. VSS score is an assessment of scar severity. Four characteristics of the scar are assessed. These are: vascularity, height, pliability, and pigmentation. Each characteristic is given a score, which are added together to give an overall score between 0 and 13. 0= normal; 13=severely scarred.
Time Frame: 2 months
Population: We will report the VSS median/mean score of 2 participants at 2 months after injection.
  The initial plan was to recruit 40 participants and follow-up with them up to 6 months; however, the study was terminated at 2 months after the recruitment of 3 subjects only due to discomfort caused by the intervention. For the VSS, only 2 out of 3 subjects completed the assessment at 2 months.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Saline Injected Half | PRP Injected Half
Number analyzed (Participants) | 2 | 2
score on a scale | 5.5 [5 to 6] | 6.5 [6 to 7]

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- PRP Injected Half: The scar to be treated will first be wiped with an alcohol swab, then measured and marked out with a marking pen such that the entirety of the scar will fit into a symmetric ellipse that is drawn, and the ellipse is filled entirely with the scar tissue. A ruler will be used to measure the scar in its greatest horizontal span, and the midway point will be marked with a vertical line. A coin flip will determine if the PRP injection (the experimental half) will be on the right half of the scar (as opposed to the left half). The half of the scar that will not receive PRP will be the control half.
  After finishing the VSS and POSAS, the area inside the experimental half of the ellipse will then be subdivided with a marking pen into 1cm x 1cm square boxes, with the plan of injecting 1mL PRP into each 1 square cm box at 0 months, 1 month, 4 months, and 6 months.
  Punch biopsies from each scar will be will be obtained at both six months and one year from enrollment.
Arm/Group | Saline Injected Half | PRP Injected Half
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Injected Half (N=3) | PRP Injected Half (N=3)
Painful Intervention (Surgical and medical procedures) | 3 (3) | 3 (3) — Pain associated with Sline/PRP injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03935594/Prot_SAP_001.pdf